CLINICAL TRIAL: NCT00856895
Title: Evaluation of Quality of Life Pre and Post Renal Transplant in Hispanic and Non-Hispanic Recipients
Brief Title: Quality of Life in Pre and Post Renal Transplant in Hispanic and Non-Hispanic Recipients
Acronym: QOL
Status: Active, not recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Juan Caicedo, Assistant Professor of Surgery; Directory of Hispanic Transplant Program,Division of Organ Transplantation, Dept of Surgery, Northwestern University
Other Study IDs: STU14943 (2689-001)
Record Dates: First submitted 2009-03-03; First posted 2009-03-06 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Transplant; Failure, Kidney
Keywords: Improved Life Quality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hispanic
- Non-Hispanic

SUMMARY:
The purpose of study is to measure the quality of life (QOL) of patients pre and post kidney transplant by asking them to fill out a survey. Patients will be asked to fill out the survey before transplant, 3 months post-transplant, and 1 year post-transplant to see how the transplant relates to any progression in quality of life.

QOL will be assessed to correlate the quality of life and aspects of renal function prospectively at pre and post-transplant across all ethnicities and variances of donor types at three time points. First, there will be a prospective assessment of QOL in the Hispanic and Non-Hispanic kidney recipients before and after transplant at NMH and Colombiana de Transplantes. Second, there will be an assessment of the Hispanic kidney patients that have been transplanted over the last 10 years at NMH and Colombiana de Transplantes, in a cross-sectional fashion. Third, there will be a comparison and determination of the differences in QOL in the Hispanic population before and after the Hispanic Transplant program was initiated in November 2006. Lastly, there will be an assessment of the social impact of the services that NMH's Hispanic Transplant Program provides to patients.

The questionnaires completed by the subjects at NMH will be the same questionnaires completed by the subjects in Colombia. The data obtained from Colombiana de Transplantes will be de-identified data and provided to us via a password protected excel file delivered to the principal investigator electronically.

DETAILED DESCRIPTION:
AIM 1: To evaluate the Quality of life in Hispanic and Non-Hispanic Kidney transplant recipients in a prospective longitudinal study using QOL questionnaires before and after the transplant. We propose to perform a prospective evaluation of QOL using the KDQOL-SF in every kidney recipient that is going to be transplanted at NMH. In addition to parameters included in the QOL instrument, we will consider ethnic background, renal function at the time of the evaluation and type of donor (deceased vs. living donor, expanded criteria donor vs. standard criteria donor), all of which has implications for the medical outcome of the transplant. An enrollment for Northwestern University is set at 750 subjects with a total approved enrollment for both sites of 1200 subjects. We plan to perform three assessments: the first before transplant, the second three months after transplant, and the third at the one year anniversary of the transplant. These milestones coincide with standard of care medical visits to the transplant center at NMH. This prospective study is going to start after the initiation of the Hispanic Kidney Transplant Program.

AIM 2: To evaluate long term QOL in Hispanic kidney transplant recipients in a cross-sectional study of NMH patients from the last 10 years using QOL questionnaires. We propose to enroll an equal number of Hispanic kidney recipients and Non-Hispanic kidney recipients transplanted over the last 10 years. We will use the KDQOL-SF to assess the current QOL in three groups according to the era of kidney transplantation: 1) Less than 1 year after transplant 2) 1-5 years after transplant and 3) 5 to 10 years post-transplant. In addition to the KDQOL-SF, we will examine their current level of renal function and the type of donor as was mention in the prospective part of this proposal.

AIM 3: To determine differences in QOL in Hispanic kidney transplant recipients before and after the Hispanic transplant program at NMH was developed.

In this specific aim, we will test the hypothesis that the cultural and educational oriented approach through the Hispanic transplant program will improve the QOL of Hispanic kidney transplant recipients and minimize differences compared to Non-Hispanic kidney recipients. To achieve this we will compare information from the cross-sectional evaluation in Aim 2 and the prospective evaluation in Aim 1 providing information before and after the inception of the Hispanic transplant program.

AIM 4: To Evaluate the social impact that the services of the NMH Hispanic Transplant program provides to the patients that participate in it. Subjects will be given a survey to complete about their experience and/or asked to participate in an interview about their experience with Northwestern Memorial's Transplant Program. If subject has participated or received a transplant and is no longer at Northwestern Memorial, a survey and letter asking for their participation may be mailed to their residence. All names will be kept confidential. Expected duration of subject participation is either a survey (15-20 min) or an interview (up to 1 hour).

ELIGIBILITY:
Inclusion Criteria:

* Pre or post renal transplant recipients ≥ 18 years of age
* Male or female
* Receiving medical care at Northwestern Memorial Hospital
* Able to read, understand and have the ability to sign the consent form and authorization for research

Exclusion Criteria:

* Pre or post renal transplant recipients < 18 years of age
* Received transplant outside of Northwestern Memorial Hospital
* Those unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 1779 kidney transplants have been performed in the last 10 years in NMH, and 220 of those kidney transplants were done in Hispanics recipients. Informed consent will be required to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2007-10; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the QOL in Hispanic and non-Hispanic Kidney Transplant Recipients | Oct. 2007 - December 2015
  To evaluate long term QOL outcomes in Hispanic and Non-Hispanic kidney transplant recipients in a prospective longitudinal study using QOL questionnaires before and after transplant.

SECONDARY OUTCOMES:
Evaluate Long Term QOL Outcomes in Hispanic and Non-Hispanic Kidney Transplant Recipients | Oct. 2007 - December 2015
  To evaluate long term QOL outcomes in Hispanic and Non-hispanic kidney transplant recipients in a cross-sectional study of Northwestern Memorial Hospital patients from the last 10 years using QOL questionnaires.

OTHER OUTCOMES:
To determine the differences in QOL outcomes in Hispanic and Non-Hispanic kidney transplant recipients | Oct. 2007 - December 2015
  To determine the differences in QOL outcomes in Hispanic kidney transplant recipients before and after recently implemented Hispanic transplant program was developed.
To Assess the social impact that services that Northwestern Memorial Hospital's Hispanic Transplant Program | Oct. 2007 - December 2015
  To Assess the social impact that services that Northwestern Memorial Hospital's Hispanic Transplant Program provides to its patients.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Caicedo, MD, Principal Investigator — Northwestern University, Northwestern Memorial Hospital
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States